CLINICAL TRIAL: NCT00505752
Title: A Phase II, Multicenter, Randomized, Assessor-blinded, Active-comparator, Dose-finding Study to Evaluate AS900672 Enriched Versus Follitropin Alfa (Gonal-f®) in Stimulating Multiple Follicular Development in Infertile Women Undergoing Assisted Reproductive Technology (ART)
Brief Title: Investigation of a Long-Acting Follicle Stimulating Hormone in Infertile Women Undergoing Assisted Reproductive Technology (ART)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27591
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Results first posted 2013-07-24 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Infertility
Keywords: Assisted reproductive technology, follicle stimulating hormone
MeSH Terms: conditions — Infertility | interventions — follitropin alfa; Follicle Stimulating Hormone; Chorionic Gonadotropin; Ovidrel

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (4):
- AS900672-Enriched 50 mcg (Experimental)
  Interventions: Drug: AS900672-Enriched 50 microgram (mcg); Drug: Follitropin alfa 150 international unit (IU); Drug: Recombinant human chorionic gonadotropin (r-hCG)
- AS900672-Enriched 100 mcg (Experimental)
  Interventions: Drug: AS900672-Enriched 100 mcg; Drug: Follitropin alfa 150 international unit (IU); Drug: Recombinant human chorionic gonadotropin (r-hCG)
- AS900672-Enriched 150 mcg (Experimental)
  Interventions: Drug: AS900672-Enriched 150 mcg; Drug: Follitropin alfa 150 international unit (IU); Drug: Recombinant human chorionic gonadotropin (r-hCG)
- Follitropin alfa 150 IU (Active Comparator)
  Interventions: Drug: Follitropin alfa 150 international unit (IU); Drug: Recombinant human chorionic gonadotropin (r-hCG)

INTERVENTIONS:
Drug: AS900672-Enriched 50 microgram (mcg) — Single injection of AS900672-Enriched (hyperglycosylated recombinant human follicle stimulating hormone [r-hFSH]), 50 mcg will be administered subcutaneously on Stimulation Day 1 (S1). Duration of treatment cycle will be up to adequate follicular response or maximum of 21 days.
  Other Names: Hyperglycosylated r-hFSH
  Arms: AS900672-Enriched 50 mcg
Drug: AS900672-Enriched 100 mcg — Single injection of AS900672-Enriched (hyperglycosylated r-hFSH), 100 mcg will be administered subcutaneously on S1. Duration of treatment cycle will up to adequate follicular response or maximum of 21 days.
  Other Names: Hyperglycosylated r-hFSH
  Arms: AS900672-Enriched 100 mcg
Drug: AS900672-Enriched 150 mcg — Single injection of AS900672-Enriched (hyperglycosylated r-hFSH), 150 mcg will be administered subcutaneously on S1. Duration of treatment cycle will up to adequate follicular response or maximum of 21 days.
  Other Names: Hyperglycosylated r-hFSH
  Arms: AS900672-Enriched 150 mcg
Drug: Follitropin alfa 150 international unit (IU) — Follitropin alfa (Gonal-f®) 150 IU will be administered subcutaneously once daily from S1 up to Stimulation Day 21 (S21) based upon ovarian response, until recombinant human chorionic gonadotropin (r-hCG) administration day. Subjects who will be receiving AS900672-Enriched 50, 100 and 150 mcg will also receive daily dose of follitropin alfa 150 IU subcutaneously from Stimulation Day 6 (S6) up to S21. Duration of treatment cycle will be up to adequate follicular response or maximum of 21 days.
  Other Names: Gonal-f®; Follicle stimulating hormone (FSH)
Drug: Recombinant human chorionic gonadotropin (r-hCG) — Recombinant human chorionic gonadotropin (r-hCG) will be administered as a single dose of 250 mcg subcutaneously, when follicular response is adequate (that is, at least 1 follicle with a diameter of greater than or equal to [>=] 18 millimeter [mm], two or more additional follicles with a diameter of >= 16 mm, and Estradiol [E2] levels will approximately 150 picogram per milliliter [pg/mL] per mature follicle).
  Other Names: Ovidrel®; Choriogonadotropin alfa

SUMMARY:
This is a Phase 2, interventional, prospective, multi-center, randomized, assessor-blind, active-comparator, dose-finding study to evaluate a new investigational long-acting follicle stimulating hormone (FSH) in infertile women who are undergoing an assisted reproductive technology (ART) procedure (In vitro fertilization/Intra cytoplasmic sperm injection [IVF/ICSI]). This study will compare 3 doses of the investigational drug versus a currently marketed drug follitropin alfa (Gonal-f® revised formulation female [RFF] Pen) in regards to the number of fertilized oocytes.

DETAILED DESCRIPTION:
Infertile women who are candidates for ART will be prospectively screened for enrollment at 24 clinical trial sites in the United States and Argentina. Enrolled subjects will start treatment using oral contraceptives (OCP) and will then receive a Gonadotropin releasing hormone (GnRH)-agonist (leuprolide acetate) for pituitary desensitization. Once down-regulation is achieved, the subjects will be randomized in a 1:1:1:1 ratio to begin ovarian stimulation with one of 3 doses of AS900672-Enriched or with follitropin alfa (Gonal-f®) daily injections. Subjects will be recruited to the four study arms in parallel. Beginning on S1, the subjects will receive either a single injection of AS900672-Enriched or start daily injections of follitropin alfa. The subjects' response to treatment will be monitored by ovarian ultrasound and E2 levels. On S6, subjects randomized to AS900672-Enriched may begin receiving supplemental follitropin alfa 150 IU, according to the each subject's ovarian response, and subjects randomized to follitropin alfa 150 IU daily injections will continue treatment at the same dose. Recombinant human chorionic gonadotropin (r-hCG, Ovidrel®) will be administered to subjects meeting response criteria and who are not at risk for ovarian hyperstimulation syndrome (OHSS). Oocyte retrieval will occur within 34-38 hours after r-hCG administration and subjects will begin luteal phase support using vaginal progesterone (Crinone® 8 percent or Prochieve® 8 percent) the following day. Fertilization will be done by conventional IVF or ICSI. Embryo transfer will occur in accordance with the specific requirements of each subject and the clinical trial site's standard practice, with the exception that a maximum of two embryos at the cleavage or blastocyst stage may be transferred. Subjects who undergo embryo transfer will be assessed for pregnancy and a follow-up visit will be performed 15-20 days post r-hCG administration. Subjects with a positive pregnancy test will undergo a confirmatory ultrasound evaluation at Day 35 - 42 post r-hCG. Additionally, all subjects recruited at certain trial centers will participate in a pharmacokinetic (PK) sub-study.

ELIGIBILITY:
Inclusion Criteria :

* Infertility and desire to conceive, justifying ART treatment
* Age between 18 and 36 years, inclusive, at time of informed consent
* Body mass index (BMI) 18 to 30 kilogram per square meter (kg/m^2), inclusive
* Regular spontaneous menstrual cycles of 21 to 35 days
* Presence of both ovaries
* Transvaginal ultrasound within 6 weeks and hysterosalpingogram, hysterosonogram or hysteroscopy within 2 years prior to beginning OCP treatment, showing no clinically significant uterine abnormality, which, in the Investigator's opinion, could impair embryo implantation or pregnancy continuation
* Normal early follicular phase (Day 2-4) serum FSH level, according to the local laboratory
* Normal serum thyroid stimulating hormone (TSH) level, according to the local laboratory
* Papanicolaou (PAP) smear test without clinically significant abnormalities within the last 6 months prior to beginning oral contraceptive therapy,
* Negative pregnancy test prior to beginning GnRH-agonist therapy
* Male partner with semen analysis which is at least adequate for ICSI within last 6 months prior to beginning GnRH agonist therapy, according to local laboratory
* Willing and able to comply with the protocol
* Voluntary provision of written informed consent, prior to any study-related procedure that was not part of normal medical care, with the understanding that the subject could withdraw consent at any time without prejudice to her future medical care, and
* Willingness to provide follow-up information on babies born as part of this study
* For subjects recruited at PK sub-study centers, voluntary provision of written informed consent to participate in the PK sub-study

Exclusion Criteria:

* Subject who require a starting dose of FSH greater than (>) 150 international unit per day (IU/day), in the opinion of the Investigator
* Screening ultrasound demonstrating more than 12 follicles less than (<) 11 mm mean diameter in either ovary
* Two or more previous ART cycles (consecutive or not) with poor response to gonadotrophin, defined as less than or equal to (=<)3 oocytes retrieved
* Three or more previous consecutive ART cycles without a biochemical or clinical pregnancy
* Previous failure of fertilization with ICSI
* A previous ART attempt in which there were no adequate or motile sperm before or after the processing of ejaculated sperm
* Previous severe OHSS
* History or presence of tumors of the hypothalamus or pituitary gland
* History or presence of ovarian, uterine or mammary cancer
* History or presence of ovarian enlargement or cyst of unknown etiology, or presence of ovarian cyst >25 mm on the day of randomization
* Presence of endometriosis Grade III - IV
* Presence of uni- or bilateral hydrosalpinx
* Abnormal gynecological bleeding of undetermined origin
* Contraindication to being pregnant and/or carrying a pregnancy to term
* History of >= 3 clinical or preclinical (absence of gestational sac) miscarriages due to any cause
* Extra-uterine pregnancy within the 3 months prior to randomization
* Clinically significant concurrent disease that would have compromised subject safety or interfered with the study assessments
* Known infection with human immunodeficiency virus (HIV), hepatitis B or C virus in the female or male partner
* Known allergy or hypersensitivity to human gonadotrophin preparations or to compounds that are structurally similar to any of the other medications administered during the study
* Any medical condition, which in the judgment of the Investigator may have interfere with the absorption, distribution, metabolism or excretion of r-hFSH
* Any active substance abuse or history of drug, medication or alcohol abuse within 5 years before screening
* ART cycle and/or ovarian stimulation within 30 days prior to informed consent
* Entered previously into this study or simultaneous participation in another clinical trial
* Subject is a smoker consuming more than 5 cigarettes per day
* In the opinion of the Investigator, either assisted hatching or pre-implantation genetic diagnosis is indicated for the subject
* Planning to undergo experimental procedures such as blastomere biopsy, or
* Any known autoimmune disease

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 520 (Actual)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zourab Bebia, MD, Study Director — EMD Serono
Locations (1):
- Local US Medical Information Office, Rockland, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- AS900672-Enriched 50 Mcg: Single injection of AS900672-Enriched (hyperglycosylated recombinant human follicle stimulating hormone [r-hFSH]), 50 microgram (mcg) administered subcutaneously on Stimulation day 1 (S1) followed by a daily dose of follitropin alfa 150 international unit (IU) subcutaneously starting from Stimulation Day 6 (S6) up to Stimulation Day 21 (S21) based upon ovarian response, until recombinant human chorionic gonadotropin (r-hCG, Ovidrel®) administration day. When follicular response was adequate (that is, at least 1 follicle with a diameter of greater than or equal to [>=] 18 millimeter [mm], two or more additional follicles with a diameter of >= 16 mm, and Estradiol [E2] levels were approximately 150 picogram per milliliter [pg/mL] per mature follicle), ovulation was triggered by single 250 mcg subcutaneous r-hCG injection. Duration of treatment cycle was up to adequate follicular response or maximum of 21 days.
- AS900672-Enriched 100 Microgram (Mcg): Single injection of AS900672-Enriched (hyperglycosylated r-hFSH), 100 mcg administered subcutaneously on S1 followed by a daily dose of follitropin alfa 150 IU subcutaneously starting from S6 up to S21 based upon ovarian response, until r-hCG administration day. When follicular response was adequate (that is, at least 1 follicle with a diameter of >= 18 mm, two or more additional follicles with a diameter of >= 16 mm, and E2 levels were approximately 150 pg/mL per mature follicle), ovulation was triggered by single 250 mcg subcutaneous r-hCG injection. Duration of treatment cycle was up to adequate follicular response or maximum of 21 days.
- AS900672-Enriched 150 Microgram (Mcg): Single injection of AS900672-Enriched (hyperglycosylated r-hFSH), 150 mcg administered subcutaneously on S1 followed by a daily dose of follitropin alfa 150 IU subcutaneously starting from S6 up to S21 based upon ovarian response, until r-hCG administration day. When follicular response was adequate (that is, at least 1 follicle with a diameter of >= 18 mm, two or more additional follicles with a diameter of >= 16 mm, and E2 levels were approximately 150 pg/mL per mature follicle), ovulation was triggered by single 250 mcg subcutaneous r-hCG injection. Duration of treatment cycle was up to adequate follicular response or maximum of 21 days.
- Follitropin Alfa 150 IU: Follitropin alfa (Gonal-f®) 150 IU administered subcutaneously once daily from S1 up to S21 based upon ovarian response, until r-hCG administration day. When follicular response was adequate (that is, at least 1 follicle with a diameter of >= 18 mm, two or more additional follicles with a diameter of >= 16 mm, and E2 levels were approximately 150 pg/mL per mature follicle), ovulation was triggered by single 250 mcg subcutaneous r-hCG injection. Duration of treatment cycle was up to adequate follicular response or maximum of 21 days.
Period: Overall Study
Arm/Group | AS900672-Enriched 50 Mcg | AS900672-Enriched 100 Microgram (Mcg) | AS900672-Enriched 150 Microgram (Mcg) | Follitropin Alfa 150 IU
Started | 132 | 128 | 128 | 132
Completed | 126 | 119 | 120 | 126
Not Completed | 6 | 9 | 8 | 6
Not completed — Adverse Event | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Lack of ovarian response | 1 | 3 | 0 | 0
Not completed — Ovarian hyperstimulation syndrome risk | 1 | 1 | 3 | 1
Not completed — No oocytes retrieved | 0 | 2 | 0 | 1
Not completed — No Fertilization | 1 | 1 | 2 | 1
Not completed — All embryos/blastocysts discarded | 0 | 0 | 1 | 1
Not completed — Other | 1 | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AS900672-Enriched 50 Mcg | AS900672-Enriched 100 Microgram (Mcg) | AS900672-Enriched 150 Microgram (Mcg) | Follitropin Alfa 150 IU | Total
Number analyzed (Participants) | 132 | 128 | 128 | 132 | 520
Age, Continuous [Median (Full Range); unit: years] | 32.0 [22 to 36] | 32.0 [22 to 36] | 32.0 [21.0 to 38] | 32.0 [24 to 36] | 32.0 [21 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 128 | 128 | 132 | 520
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Fertilized Oocytes (2 Pronuclei [PN])
Description: Oocytes were fertilized using Intra-cytoplasmic Sperm Injection (ICSI) technique which is an in-vitro fertilization procedure in which a single sperm is injected directly into an egg under a microscope. The appearance of 2PN is the first sign of successful fertilization as observed during in vitro fertilization, and is usually observed after ICSI. The zygote is then termed 2PN.
Time Frame: Ovum pick-up (OPU) day (34-38 hours post r-hCG administration day [end of stimulation cycle {approximately 21 days}])
Population: Intention-to-treat (ITT) population included all the participants who were randomized to study treatment. 'N' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: 2PN oocytes
Arm/Group | AS900672-Enriched 50 Mcg | AS900672-Enriched 100 Microgram (Mcg) | AS900672-Enriched 150 Microgram (Mcg) | Follitropin Alfa 150 IU
Number analyzed (Participants) | 130 | 122 | 124 | 131
2PN oocytes | 7.0 (4.7) | 8.7 (4.9) | 9.2 (6.0) | 6.7 (4.2)

2. Secondary Outcome: Percentage of Participants With Clinical Pregnancy
Description: Clinical pregnancy was defined as the presence of one or more fetal sacs with fetal heart activity on the Day 35-42 post r-hCG ultrasound examination.
Time Frame: Day 35-42 post r-hCG administration day (end of stimulation cycle [approximately 21 days])
Population: ITT population included all the participants who were randomized to study treatment. 'N' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: Percentage of participants
Arm/Group | AS900672-Enriched 50 Mcg | AS900672-Enriched 100 Microgram (Mcg) | AS900672-Enriched 150 Microgram (Mcg) | Follitropin Alfa 150 IU
Number analyzed (Participants) | 128 | 120 | 122 | 128
Percentage of participants | 39.1 | 40.8 | 35.2 | 43.8

ADVERSE EVENTS:
Time Frame: Stimulation Day 1 (S1) up to Day 35-42 post r-hCG administration day (end of stimulation cycle [approximately 21 days])
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an investigational medicinal product (IMP), regardless of causal relationship and even if no IMP has been administered.
Arm/Group | AS900672-Enriched 50 Mcg | AS900672-Enriched 100 Microgram (Mcg) | AS900672-Enriched 150 Microgram (Mcg) | Follitropin Alfa 150 IU
Serious Adverse Events (participants affected / at risk) | 5/132 | 5/128 | 4/128 | 6/132
Other Adverse Events (participants affected / at risk) | 90/132 | 85/128 | 84/128 | 82/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AS900672-Enriched 50 Mcg (N=132) | AS900672-Enriched 100 Microgram (Mcg) (N=128) | AS900672-Enriched 150 Microgram (Mcg) (N=128) | Follitropin Alfa 150 IU (N=132)
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Heterotopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 2 | 0
Ovarian Hyperstimulation Syndrome (Reproductive system and breast disorders) | 0 | 1 | 1 | 1
Ovarian torsion (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Umbilical cord abnormality (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Ventriculo septal defect (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Heart disease congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AS900672-Enriched 50 Mcg (N=132) | AS900672-Enriched 100 Microgram (Mcg) (N=128) | AS900672-Enriched 150 Microgram (Mcg) (N=128) | Follitropin Alfa 150 IU (N=132)
Procedural pain (Injury, poisoning and procedural complications) | 35 | 29 | 27 | 39
Headache (Nervous system disorders) | 23 | 22 | 22 | 28
Abdominal distension (Gastrointestinal disorders) | 15 | 16 | 22 | 22
Adnexa uteri pain (Reproductive system and breast disorders) | 20 | 14 | 14 | 15
Nausea (Gastrointestinal disorders) | 11 | 10 | 12 | 16
Uterine spasm (Reproductive system and breast disorders) | 3 | 7 | 11 | 5
Fatigue (General disorders) | 5 | 4 | 4 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 8 | 4 | 4
Constipation (Gastrointestinal disorders) | 3 | 5 | 7 | 3
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 6 | 5 | 10 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other